CLINICAL TRIAL: NCT03821935
Title: A Phase 1 First-in Human, Multi-Center, Open Label Dose-Escalation Study to Determine the Safety, Tolerability, Pharmacokinetics and RP2D of Livmoniplimab (ABBV-151) as a Single Agent and in Combination With Budigalimab (ABBV-181) in Subjects With Locally Advanced or Metastatic Solid Tumors
Brief Title: Study to Determine the Safety, Tolerability, Pharmacokinetics and Recommended Phase 2 Dose (RP2D) of Livmoniplimab (ABBV-151) as a Single Agent and in Combination With Budigalimab (ABBV-181) in Participants With Locally Advanced or Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M19-345; 2023-508281-15-00 (Other: EU CT)
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumors Cancer
Keywords: Advanced Solid Tumors Cancer; cancer; Solid Tumors; metastatic; monotherapy; combination therapy; triple negative breast cancer (TNBC); pancreatic adenocarcinoma; urothelial cancer; hepatocellular carcinoma (HCC); head and neck squamous cell carcinoma (HNSCC); Colorectal cancer; Ovarian granulosa cell tumors
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Triple Negative Breast Neoplasms; Carcinoma, Hepatocellular; Squamous Cell Carcinoma of Head and Neck; Colorectal Neoplasms | interventions — budigalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (15):
- Dose Escalation: Cohort 1 Livmoniplimab (Experimental): Various doses of Livmoniplimab administered during dose escalation to determine the Recommended Phase 2 Dose (RP2D).
  Interventions: Drug: Livmoniplimab
- Dose Escalation: Cohort 2 Livmoniplimab + Budigalimab (Experimental): Various doses of Livmoniplimab + Budigalimab administered during dose escalation to determine the Recommended Phase 2 Dose (RP2D).
  Interventions: Drug: Livmoniplimab; Drug: Budigalimab
- Dose Expansion: Cohort 3 Livmoniplimab + Budigalimab (Experimental): Participants with programmed cell death protein 1 (PD-1)-naïve pancreatic adenocarcinoma will receive livmoniplimab at the RP2D Q2W plus budigalimab Dose A administered Q4W.
  Interventions: Drug: Livmoniplimab; Drug: Budigalimab
- Dose Expansion: Cohort 4 Livmoniplimab + Budigalimab (Experimental): Participants with PD-1-ref urothelial cancer will receive livmoniplimab at the RP2D Q2W plus budigalimab Dose A administered Q4W.
  Interventions: Drug: Livmoniplimab; Drug: Budigalimab
- Dose Expansion: Cohort 5 Livmoniplimab + Budigalimab (Experimental): Participants with PD-1-naïve hepatocellular carcinoma (HCC) will receive livmoniplimab at the RP2D Q2W plus budigalimab Dose A administered Q4W.
  Interventions: Drug: Livmoniplimab; Drug: Budigalimab
- Dose Expansion: Cohort 6 Livmoniplimab + Budigalimab (Experimental): Participants with PD-1-ref head and neck squamous cell carcinoma (HNSCC) will receive livmoniplimab at the RP2D Q2W plus budigalimab Dose A administered Q4W.
  Interventions: Drug: Livmoniplimab; Drug: Budigalimab
- Dose Expansion: Cohort 7 Livmoniplimab + Budigalimab (Experimental): Participants with PD-1-naïve microsatellite stable colorectal cancer (MSS-CRC) [unselected] will receive livmoniplimab at the RP2D Q2W plus budigalimab Dose A administered Q4W.
  Interventions: Drug: Livmoniplimab; Drug: Budigalimab
- Dose Expansion: Cohort 8 Livmoniplimab + Budigalimab (Experimental): Participants with non-small cell lung cancer (NSCLC) [programmed death ligand 1 (PDL1) relapsed/refractory (R/R)] will receive livmoniplimab at the RP2D Q2W plus budigalimab Dose A administered Q4W.
  Interventions: Drug: Livmoniplimab; Drug: Budigalimab
- Dose Expansion: Cohort 10A Livmoniplimab + Budigalimab (Experimental): Participants with microsatellite stable colorectal cancer (MSS-CRC) [consensus molecular subtype 4 (CMS4) enriched] will receive livmoniplimab at the dose B Q3W plus budigalimab Dose B administered Q3W.
  Interventions: Drug: Livmoniplimab; Drug: Budigalimab
- Dose Expansion: Cohort 10B Livmoniplimab + Budigalimab (Experimental): Participants with MSS-CRC (CMS4 enriched) will receive livmoniplimab at the dose C Q3W plus budigalimab Dose B administered Q3W.
  Interventions: Drug: Livmoniplimab; Drug: Budigalimab
- Dose Expansion: Cohort 11A Livmoniplimab + Budigalimab (Experimental): Participants with PD-1-ref urothelial cancer will receive livmoniplimab at the Dose B Q3W plus budigalimab Dose B administered Q3W.
  Interventions: Drug: Livmoniplimab; Drug: Budigalimab
- Dose Expansion: Cohort 11B Livmoniplimab + Budigalimab (Experimental): Participants with PD-1-ref urothelial cancer will receive livmoniplimab at the Dose C Q3W plus budigalimab Dose B administered Q3W.
  Interventions: Drug: Livmoniplimab; Drug: Budigalimab
- Dose Expansion: Cohort 11C Budigalimab (Experimental): Participants with PD-1-ref urothelial cancer will receive budigalimab Dose B administered Q3W.
  Interventions: Drug: Budigalimab
- Dose Expansion: Cohort 12A Livmoniplimab + Budigalimab (Experimental): Participants with PD-1-naïve ovarian granulosa (OG) cell tumors will receive livmoniplimab at the Dose B Q3W plus budigalimab Dose B administered Q3W.
  Interventions: Drug: Livmoniplimab; Drug: Budigalimab
- Dose Expansion: Cohort 12B Livmoniplimab + Budigalimab (Experimental): Participants with PD-1-naïve ovarian granulosa (OG) cell tumors will receive livmoniplimab at the Dose C Q3W plus budigalimab Dose B administered Q3W.
  Interventions: Drug: Livmoniplimab; Drug: Budigalimab

INTERVENTIONS:
Drug: Livmoniplimab — Liquid for intravenous infusion.
  Other Names: ABBV-151
  Arms: Dose Escalation: Cohort 1 Livmoniplimab; Dose Escalation: Cohort 2 Livmoniplimab + Budigalimab; Dose Expansion: Cohort 10A Livmoniplimab + Budigalimab; Dose Expansion: Cohort 10B Livmoniplimab + Budigalimab; Dose Expansion: Cohort 11A Livmoniplimab + Budigalimab; Dose Expansion: Cohort 11B Livmoniplimab + Budigalimab; Dose Expansion: Cohort 12A Livmoniplimab + Budigalimab; Dose Expansion: Cohort 12B Livmoniplimab + Budigalimab; Dose Expansion: Cohort 3 Livmoniplimab + Budigalimab; Dose Expansion: Cohort 4 Livmoniplimab + Budigalimab; Dose Expansion: Cohort 5 Livmoniplimab + Budigalimab; Dose Expansion: Cohort 6 Livmoniplimab + Budigalimab; Dose Expansion: Cohort 7 Livmoniplimab + Budigalimab; Dose Expansion: Cohort 8 Livmoniplimab + Budigalimab
Drug: Budigalimab — Lyophilized powder for solution for intravenous infusion.
  Other Names: ABBV-181
  Arms: Dose Escalation: Cohort 2 Livmoniplimab + Budigalimab; Dose Expansion: Cohort 10A Livmoniplimab + Budigalimab; Dose Expansion: Cohort 10B Livmoniplimab + Budigalimab; Dose Expansion: Cohort 11A Livmoniplimab + Budigalimab; Dose Expansion: Cohort 11B Livmoniplimab + Budigalimab; Dose Expansion: Cohort 11C Budigalimab; Dose Expansion: Cohort 12A Livmoniplimab + Budigalimab; Dose Expansion: Cohort 12B Livmoniplimab + Budigalimab; Dose Expansion: Cohort 3 Livmoniplimab + Budigalimab; Dose Expansion: Cohort 4 Livmoniplimab + Budigalimab; Dose Expansion: Cohort 5 Livmoniplimab + Budigalimab; Dose Expansion: Cohort 6 Livmoniplimab + Budigalimab; Dose Expansion: Cohort 7 Livmoniplimab + Budigalimab; Dose Expansion: Cohort 8 Livmoniplimab + Budigalimab

SUMMARY:
The study will determine the recommended Phase 2 dose (RP2D) of livmoniplimab (ABBV-151) administered as monotherapy and in combination with budigalimab (ABBV-181) as well as to assess the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of livmoniplimab alone and in combination with budigalimab. The study will consist of 2 parts: dose escalation and dose expansion.

ELIGIBILITY:
Inclusion Criteria:

* For Dose Escalation only: Participants with an advanced solid tumor who are considered refractory to or intolerant of all existing therapy(ies) known to provide a clinical benefit for their condition. Additionally, participants who have been offered standard therapies and refused, or who are considered ineligible for standard therapies, may be eligible for this study on a case-by-case basis, after discussion with and agreement from the sponsor. Participants with pancreatic adenocarcinoma, urothelial cancer (UC), hepatocellular carcinoma (HCC), or head and neck squamous cell carcinoma (HNSCC) who are being considered for the dose escalation cohorts must also meet the histology specific eligibility criteria described below for dose expansion.
* For Dose Expansion only participants must meet criteria specific to the type of cancer:

  * Pancreatic adenocarcinoma and have disease progression during or after 1 systemic therapy (gemcitabine monotherapy or in combination with other agents, FOLFIRINOX [or another regimen including both 5-fluorouracil and oxaliplatin], capecitabine monotherapy or in combination with other agents) administered in the adjuvant, locally advanced, or metastatic setting. If the therapy was used in an adjuvant setting, disease progression must have occurred within 6 months of completing adjuvant therapy.
  * UC of the bladder and urinary tract and must have progressed following treatment with:
  * Cohort 4: A platinum-based regimen (administered in any line of therapy) and a programmed death 1/programmed death ligand 1 (PD1/PDL1) antagonist administered in the recurrent or metastatic setting (progression following a PD1/PDL1 antagonist is defined as unequivocal progression on or within 3 months of the last dose of anti-PD1 or anti-PDL1 therapy).
  * Cohort 11: One or more prior line of therapy in the locally advanced or metastatic setting. Participant must have experienced radiographic progression or relapse during or after a CPI (anti-PD1 or anti-PD-L1) for locally advanced or metastatic disease.
  * HCC and must have disease progression during or after 1 prior line of systemic therapy.
  * HNSCC (arising from the oral cavity, oropharynx, hypopharynx, or larynx) and must have progressed following treatment with platinum-based regimen (administered in any line of therapy) and a PD1/PDL1 antagonist administered in the recurrent or metastatic setting (progression following a PD1/PDL1 antagonist is defined as unequivocal progression on or within 3 months of the last dose of anti-PD1 or anti-PDL1 therapy).
  * Microsatellite stable colorectal cancer (MSS-CRC) [unselected] participants with microsatellite stable or mismatch repair proficient colorectal adenocarcinoma (as determined by polymerase chain reaction (PCR)/Next-Generation sequencing (NGS) or immunohistochemistry (IHC), respectively) who have received 1-2 prior chemotherapy regimens.
  * Non-small cell lung cancer (NSCLC) relapsed/refractory (R/R): Participants with histologically or cytologically confirmed advanced or metastatic NSCLC who have received 1 prior line of chemotherapy and 1 prior anti-PD-(L)1 antibody, administered either concurrently or sequentially in the metastatic setting.
  * MSS-CRC (CMS4 enriched): Participants with microsatellite stable or mismatch repair proficient colorectal adenocarcinoma who have received prior fluorouracil-based combination chemotherapy regimens including oxaliplatin and irinotecan (with or without VEGF and/or EGFR targeted agents) and with a CMS4 subtype as determined by NGS of tumor biopsies. Archival tissue must be submitted for assessment of CMS4 subtype status during prescreening. Participants must have progressed on or refused available standard of care therapies. Additionally, participant who are considered not appropriate or ineligible for available standard of care therapies per investigator assessment will be eligible for this study.
  * Ovarian granulosa (OG) cell tumor: Participants with histologically confirmed advanced nonresectable or metastatic adult granulosa cell tumor of the ovary that is not amenable to curative intent surgery or radiation. Additionally, there is documentation of radiological evidence of relapse after at least 1 line of systemic chemotherapy.
* Participant has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1.
* Participant has adequate bone marrow, renal, hepatic, and coagulation function.
* Must have a viral status consistent with the requirements described in the protocol specific to type of cancer and stage of study (Dose Escalation or Dose Expansion).

Exclusion Criteria:

* For Dose Expansion only:

  * Participants with HCC, pancreatic adenocarcinoma, or MSS-CRC having prior exposure to a prior PD-1/PD-L1 antagonist in any line of therapy.
  * Participants (except for participants with urothelial cancer or HNSCC) who have had prior exposure to immunotherapies as listed in the protocol.
* Has received anticancer therapy including chemotherapy, immunotherapy, radiation therapy, biologic, herbal therapy, or any investigational therapy within a period of 5 half-lives or 28 days (whichever is shorter), prior to the first dose of the study drug.
* Participant has unresolved AEs > Grade 1 from prior anticancer therapy except for alopecia.
* Has a history of primary immunodeficiency, bone marrow transplantation, solid organ transplantation, or previous clinical diagnosis of tuberculosis.
* Has a known uncontrolled metastases to the central nervous system (with certain exceptions).
* Current or prior use of immunosuppressive medication within 14 days prior to the first dose of the study drug.
* Has clinically significant uncontrolled condition(s).
* History of inflammatory bowel disease, interstitial lung disease or pneumonitis, myocarditis, Stevens-Johnson syndrome, toxic epidermal necrolysis or drug reaction with eosinophilia and systemic symptoms (DRESS).
* Live vaccine administration <= 28 days prior to the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation: Recommended Phase 2 Dose (RP2D) Livmoniplimab Monotherapy | Up to 28 days after the first dose of Livmoniplimab monotherapy
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for the dose expansion arms, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation portion of the study.
Dose Escalation: RP2D Livmoniplimab + Budigalimab Combination Therapy | Up to 28 days after the first dose of Livmoniplimab and Budigalimab combination therapy
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for the dose expansion arms, based on safety, tolerability, efficacy, pharmacokinetics (PK), and pharmacodynamic (PD) data collected during the dose escalation portion of the study.
Dose Expansion: Objective Response Rate (ORR) | Up to approximately 6 months after the first dose date of last participant in Dose Expansion
  ORR defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
Dose Expansion: Duration of Response (DOR) | Up to approximately 6 months after the first dose date of last participant in Dose Expansion
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Dose Expansion: Progression-free Survival (PFS) | Up to approximately 6 months after the first dose date of last participant in Dose Expansion
  Progression-free survival is defined as the time from the participant's first dose of study treatment (livmoniplimab or budigalimab) to the first date of either disease progression or death, whichever occurs first.
Maximum Observed Serum Concentration (Cmax) of Livmoniplimab | Up to approximately 70 days after initial dose of study drug
  Maximum Serum Concentration (Cmax) of livmoniplimab.
Time to Maximum Observed Serum Concentration (Tmax) of Livmoniplimab | Up to approximately 70 days after initial dose of study drug
  Time to maximum serum concentration (Tmax) of livmoniplimab.
Area Under the Plasma Concentration-time Curve over time from 0 to last measurable concentration (AUCτ) of Livmoniplimab | Up to approximately 70 days after initial dose of study drug
  Area under the serum concentration-time curve from time 0 to the time of the last measurable concentration (AUCτ) of livmoniplimab.
Terminal-phase Elimination Rate Constant (β) of Livmoniplimab | Up to approximately 70 days after initial dose of study drug
  Apparent terminal phase elimination rate constant (β or Beta) of livmoniplimab.
Terminal Phase Elimination Half-life (t1/2) of Livmoniplimab | Up to approximately 70 days after initial dose of study drug
  Terminal phase elimination half-life (t1/2) of livmoniplimab.
Maximum Observed Serum Concentration (Cmax) of Budigalimab | Up to approximately 70 days after initial dose of study drug
  Maximum Serum Concentration (Cmax) of budigalimab.
Time to Maximum Observed Serum Concentration (Tmax) of Budigalimab | Up to approximately 70 days after initial dose of study drug
  Time to maximum serum concentration (Tmax) of budigalimab.
Area Under the Plasma Concentration-time Curve over time from 0 to last measurable concentration (AUCτ) of Budigalimab | Up to approximately 70 days after initial dose of study drug
  Area under the serum concentration-time curve from time 0 to the time of the last measurable concentration (AUCτ) of budigalimab.
Terminal-phase Elimination Rate Constant (β) of Budigalimab | Up to approximately 70 days after initial dose of study drug
  Apparent terminal phase elimination rate constant (β or Beta) of budigalimab.
Terminal Phase Elimination Half-life (t1/2) of Budigalimab | Up to approximately 70 days after initial dose of study drug
  Terminal phase elimination half-life (t1/2) of budigalimab.
Number of Participants With Adverse Events (AEs) | Up to approximately 9 months after the first dose date of last participant
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above.
Change in Vital Signs | Up to approximately 6 months after the first dose date of last participant
  Number of participants with clinically significant change from baseline in vital signs like systolic and diastolic blood pressure will be reported.
Change in Laboratory Parameters | Up to approximately 6 months after the first dose date of last participant
  Number of participants with clinically significant change from baseline in clinical laboratory test results like hematology will be reported.
Change in Electrocardiogram (ECG) | Up to approximately 6 months after the first dose date of last participant
  12-lead resting ECGs will be recorded. Parameters include RR interval, PR interval, QT interval, and QRS duration.
Incidence of Anti-drug Antibody (ADA) | Up to approximately 6 months after the first dose date of last participant
  The number of participants with anti-drug antibodies.
Dose Expansion Cohorts 10 to 12: Overall Survival (OS) | Up to approximately 6 months after the first dose date of last participant in Cohorts 10 to 12
  OS is defined as time from first study treatment to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (64):
- United States (21):
  - Highlands Oncology Group, PA /ID# 218942, Springdale, Arkansas
  - City of Hope National Medical Center /ID# 265620, Duarte, California
  - City of Hope Orange County Lennar Foundation Cancer Center /ID# 270785, Irvine, California
  - Yale University School of Medicine /ID# 208356, New Haven, Connecticut
  - AdventHealth Celebration /ID# 224860, Celebration, Florida
  - Duplicate_AdventHealth Cancer Institute - Orlando /ID# 226953, Orlando, Florida
  - Indiana Univ School Medicine /ID# 208384, Indianapolis, Indiana
  - Community Health Network, Inc. /ID# 257032, Indianapolis, Indiana
  - Univ Michigan Med Ctr /ID# 221129, Ann Arbor, Michigan
  - Washington University-School of Medicine /ID# 259684, St Louis, Missouri
  - Intermountain Health West End Clinic Gynecologic Oncology /ID# 266171, Billings, Montana
  - NYU Langone Medical Center /ID# 209822, New York, New York
  - Icahn School of Medicine at Mount Sinai /ID# 264653, New York, New York
  - Carolina BioOncology Institute /ID# 208358, Huntersville, North Carolina
  - The Ohio State University - The James /ID# 217611, Columbus, Ohio
  - Ou Health - Stephenson Cancer Center /ID# 268826, Oklahoma City, Oklahoma
  - Sarah Cannon Research Institute (SMO/Network/Consortium) /ID# 264900, Nashville, Tennessee
  - Renovatio clinical /ID# 265109, El Paso, Texas
  - NEXT Oncology /ID# 208930, San Antonio, Texas
  - Renovatio Clinical /ID# 265054, The Woodlands, Texas
  - University of Washington Medical Center /ID# 268854, Seattle, Washington
- Australia (2):
  - Chris O'Brien Lifehouse /ID# 213236, Camperdown, New South Wales
  - Icon Cancer Centre /ID# 224961, South Brisbane, Queensland
- Cliniques Universitaires UCL Saint-Luc /ID# 218466, Brussels, Brussels Capital, Belgium
- University Health Network_Princess Margaret Cancer Centre /ID# 209423, Toronto, Ontario, Canada
- France (4):
  - CHU Toulouse - Hopital Purpan /ID# 218667, Toulouse, Haute-Garonne
  - Centre Leon Berard /ID# 218515, Lyon, Rhone
  - Institut Gustave Roussy /ID# 218668, Villejuif, Val-de-Marne
  - Centre Jean Perrin /ID# 218669, Clermont-Ferrand
- Kliniken Essen-Mitte, Evangelische Huyssens-Stiftung /ID# 269587, Essen, North Rhine-Westphalia, Germany
- Israel (5):
  - Rambam Health Care Campus /ID# 222198, Haifa, H_efa
  - The Chaim Sheba Medical Center /ID# 209037, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 222199, Tel Aviv, Tel Aviv
  - Hadassah Medical Center-Hebrew University /ID# 257918, Jerusalem
  - Rabin Medical Center /ID# 258479, Petah Tikva
- Istituto Europeo Di Oncologia /Id# 266053, Milan, Milano, Italy
- Japan (3):
  - National Cancer Center Hospital East /ID# 224808, Kashiwa-shi, Chiba
  - Hyogo Cancer Center /ID# 272553, Akashi-shi, Hyōgo
  - National Cancer Center Hospital /ID# 209421, Chuo-ku, Tokyo
- Poland (3):
  - Jagiellonskie Centrum Innowacji Sp. z o.o. /ID# 266194, Krakow, Lesser Poland Voivodeship
  - Narodowy Instytut Onkologii Im. Marii Sklodowskiej-Curie Panstwowy Instytut Bada /ID# 266147, Warsaw, Masovian Voivodeship
  - Instytut Centrum Zdrowia Matki Polki /ID# 266324, Lodz, Łódź Voivodeship
- Pan American Center for Oncology Trials, LLC /ID# 217475, Rio Piedras, Puerto Rico
- South Korea (7):
  - Gachon University Gil Medical Center /ID# 257572, Incheon, Gyeonggido
  - Chonnam National University Hwasun Hospital /ID# 257573, Hwasun-gun, Jeonranamdo
  - Korea University Anam Hospital /ID# 257574, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital /ID# 218513, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 266799, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 265865, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 218512, Seoul
- Spain (8):
  - Clinica Universidad de Navarra - Pamplona /ID# 266632, Pamplona, Navarre
  - Hospital Universitari Vall d'Hebron /ID# 265290, Barcelona
  - Hospital Clinic de Barcelona /ID# 221106, Barcelona
  - Clinica Universidad de Navarra - Madrid /ID# 265299, Madrid
  - Hospital Universitario Ramón y Cajal /ID# 265298, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz /ID# 220928, Madrid
  - Hospital Universitario HM Sanchinarro /ID# 265294, Madrid
  - Hospital Clinico Universitario de Valencia /ID# 221107, Valencia
- Taiwan (6):
  - Kaohsiung Chang Gung Memorial Hospital /ID# 265560, Kaohsiung City, Kaohsiung
  - National Taiwan University Hospital /ID# 218490, Taipei City, Taipei
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 257634, Kaohsiung City
  - China Medical University Hospital /ID# 218492, Taichung
  - Taipei Veterans General Hosp /ID# 257635, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 265551, Taoyuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shimizu T, Powderly J, Abdul Razak A, LoRusso P, Miller KD, Kao S, Kongpachith S, Tribouley C, Graham M, Stoll B, Patel M, Sahtout M, Blaney M, Leibman R, Golan T, Tolcher A. First-in-human phase 1 dose-escalation results with livmoniplimab, an antibody targeting the GARP:TGF-ss1 complex, as monotherapy and in combination with the anti-PD-1 antibody budigalimab in patients with advanced solid tumors. Front Oncol. 2024 Oct 29;14:1376551. doi: 10.3389/fonc.2024.1376551. eCollection 2024. PMID 39534099
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M19-345